CLINICAL TRIAL: NCT02526576
Title: A Phase II Double-blind, Randomized, Study to Assess the Efficacy of Facial Fat Grafts Supplemented With Autologous, Adipose Derived Stromal Vascular Fraction (SVF)
Brief Title: Adipose Derived Stem Cells in Facial Fat Grafting
Acronym: SVF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antria (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSVF0002
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Facial Atrophy
Keywords: Facial Atrophy; Autologous; Adult; Adipose Derived Stem Cells; Stromal Vascular Fraction; Collagenase
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stromal Vascular Fraction (Experimental): Subjects will receive stromal vascular fraction assisted fat transfer.
  Interventions: Biological: Stromal Vasular Fraction; Procedure: Biopsy
- Biopsy for Control -regular fat transfer (Active Comparator): Subjects will receive regular fat transfer. A biopsy procedure will analyzes the different between experimental and control groups.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Biological: Stromal Vasular Fraction — The stromal vascular fraction obtained from adipose tissue will be added to the graft
  Other Names: Stromal Vascular Fraction; Adiployx
  Arms: Stromal Vascular Fraction
Procedure: Biopsy — A subgroup of each arm (2 subjects from each arm) will undergo a fat transfer behind each ear to be removed via biopsy after 12 months

SUMMARY:
This phase two, randomized, double-blind study is designed to demonstrate the enhanced efficacy of SVF-enriched autologous facial fat grafts, in relation to standard, non-SVF enriched, facial fat grafts by evaluating volumetric retention and contour of the engrafted region over the course of one year.

DETAILED DESCRIPTION:
Human Adipose Tissue is considered as a new source for Stromal Stem Cells and offers a large therapeutic potential for many rare and common diseases that impacts millions of patients worldwide. The Stromal Vascular Fraction (SVF) of Adipose Tissue is relatively easy to extract with minimally invasive procedures such as elective liposuction in large quantities and therefore may be a cost effective source for cellular therapies in a wide range of medical specialties.

The term "Facial Atrophy" describes the lost of subcutaneous fat within the face and can be a result of the aging process as well as some pathological diseases. It can be corrected via autologous fat transfer but usually the majority of the grafted cells will die after 6-12 months. Several publications demonstrate that the addition of SVF cells to the graft may enhance the graft survival.

This double blind, randomized study aims to demonstrated the efficacy of Antria Cell Preparation Process in autologous facial fat grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, Age 18 to 70 years old
2. Subjects that are eligible for liposuction and facial fat grafting procedures for cosmetic purposes and facial atrophy.
3. Subjects must require augmentation to the infra-malar region. Furthermore, facial engraftment to additional, non-study related regions is optional, but not required.
4. Inframalar Atrophy Assessment Scale of 2 to 4
5. Facial volume defect range: 2 to 10 mL
6. Body Mass Index (BMI) between and including 22 and 29
7. Able to understand and provide written and verbal informed consent
8. Fitzpatrick Scale 1 to 6

Exclusion Criteria:

1. Currently taking or have taken None Steroid Anti-inflammatory Drugs (NSAIDs) within last two weeks or corticosteroids within the last six weeks prior to screening
2. Diagnosis of any of the following medical conditions:

   * Active malignancy (diagnosed within 5 years), except for treated non-melanoma skin cancer or other non-invasive or in-situ neoplasm (e.g. cervical cancer)
   * Active infection
   * Type I or Type II Diabetes
   * Skin/Bone deformities in the face, including scaring or hyperpigmentation within the graft site.
3. Subjects who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits, dementia, and/or otherwise considered by the Investigator to be unlikely to complete the study)
4. Subjects with a known drug or alcohol dependence within the past 12 months as judged by the Investigator
5. Dermal fillers or facial reconstruction within the past 24 months, Subjects must also refrain from such procedures during the duration of the study.
6. Subjects with major illnesses involving the renal, hepatic, cardiovascular, and/or nervous systems.
7. Subjects with elevated kidney and/or liver functions
8. Any other disease condition or laboratory results that in the opinion of the investigator may be clinically significant and render the subject inappropriate for the study procedure(s), may alter the accuracy of study results, or increase risk for subjects.
9. Subjects with life-expectancies less than 9 months
10. Subjects with known collagenase allergies
11. Subjects with idiopathic or drug-induced coagulopathy
12. Pregnant females
13. On radiotherapy or chemotherapy agents
14. Taking strong CYP450 inhibitors
15. Subjects with a history of keloids or hypertrophic scar formations
16. Previous treatment with any synthetic fillers in the inframalar area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Volume retention | 12 months
  To demonstrate that SVF administration, in concert with autologous facial fat grafts, is more efficacious, with regards to graft survival, than standard, non-SVF enhanced, autologous facial fat grafts

SECONDARY OUTCOMES:
Number of Participants ith autologous facial fat grafts via laboratory results | 36 months
  To monitor the safety of SVF administration along with autologous facial fat grafts via laboratory results
Changes in the quality of skin | 12 months
  a blinded and independent investigator will assess any changes to the quality of skin

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Rahimian, MD, Study Director — Antria
Locations (1):
- Delmont Surgery Center, Delmont, Pennsylvania, United States

REFERENCES:
- [Derived] Bustos SS, Vyas K, Huang TCT, Suchyta M, LeBrasseur N, Cotofana S, Wyles SP, Mardini S. Pharmacologic and Other Noninvasive Treatments of the Aging Face: A Review of the Current Evidence. Plast Reconstr Surg. 2024 Oct 1;154(4):829e-842e. doi: 10.1097/PRS.0000000000010767. Epub 2023 May 26. PMID 39314107
- See also: Sponsor's website — http://www.antria.org
- See also: Site's website — http://artisan-plasticsurgery.com/